CLINICAL TRIAL: NCT04494594
Title: Evaluating the Efficacy of a Mobile App (Drinks:Ration) and Personalized Text and Push Messaging to Reduce Alcohol Consumption in a Veteran Population: Protocol for a Randomized Controlled Trial
Brief Title: Drinks:Ration - Combat Stress Randomized Controlled Trial
Acronym: Drinks:Ration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: University of Liverpool (Other); British Army (Unknown); Combat Stress (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HR-19/20-17438
Record Dates: First submitted 2020-07-23; First posted 2020-07-31 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2021-06

CONDITIONS: Alcohol Abuse; Mental Disorder; Mental Health Issue
Keywords: alcohol; mobile health; sms text message; push notifications
MeSH Terms: conditions — Alcoholism; Mental Disorders

STUDY DESIGN:
Intervention Model Description: This is a two-arm participant blinded (single-blinded) RCT, comparing a smartphone app (control arm) which includes feedback on baseline self-reported alcohol consumption, with a smartphone app (intervention arm) that includes individualised normative feedback, plus features designed to enhance participant motivation, app interactive feedback and self-efficacy in modifying their alcohol consumption. In this study, both the control and intervention arms will be delivered via one smartphone app known as Drinks:Ration. Participants in the control arm are given access only to alcohol consumption feedback based on publicly available health guidance and reminder messaging to consult the feedback. Those in the intervention arm are given full access to the app which includes all theoretically driven components and messaging (discussed further in Intervention section). Both arms will be asked to use the app for 28-days.
Who Masked: Participant, Care Provider
Masking Description: Randomisation occurs when a quick response (QR) code is generated and a unique proxy identifier and participant gender is assigned. At this point, participants are automatically randomised to receive the control or intervention arm and are blinded. Block randomisation, of size 2, will be used to ensure equal gender distribution across both conditions. The randomisation procedure is done automatically by the Drinks:Ration platform with no human involvement except to provide a proxy identifier and gender.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Sham Comparator)
  Interventions: Behavioral: Drinks:Ration app
- Intervention (Active Comparator)
  Interventions: Behavioral: Drinks:Ration app

INTERVENTIONS:
Behavioral: Drinks:Ration app — Drinks:Ration (www.drinksration.app; formerly called InDEx) app has been developed following the Medical Research Council Complex Intervention Guidelines and using co-design methodology by the King's Centre for Military Health Research (at King's College London) and the University of Liverpool, supported by experts in smartphone app development, epidemiology, addiction psychiatry, and military mental health. The app is designed to support veterans drinking at a hazardous or harmful level by providing detailed advice and support over a minimum of 28-day period. The app is theoretically underpinned to enhance participants motivation and self-efficacy in modifying their alcohol consumption by means of Behaviour Change Theory in the content displayed, and the messaging sent to participants.

SUMMARY:
Alcohol misuse is higher in the United Kingdom (UK) Armed Forces (AF) than the general population. Previous research has shown that interventions delivered via smartphone are efficacious in promoting self-monitoring of alcohol use, have utility in reducing alcohol consumption and have a broad reach. The main objective of this participant blinded (single-blinded) Randomised Controlled Trial (RCT) is to assess the efficacy of a 28-day brief alcohol intervention delivered via a smartphone app (Drinks:Ration) in reducing weekly self-reported alcohol consumption between baseline and 3-month follow-up among veterans who drink at a hazardous or harmful level and are receiving, or have received, support for mental health symptoms in a clinical setting.

Methods: In a two-arm single-blinded Randomised Controlled Trial (RCT), a smartphone app which includes interactive features designed to enhance participant motivation and personalised messaging is compared to a smartphone app which only provides Government guidance on alcohol consumption. The trial will be conducted in a veteran population who have sought help through Combat Stress; a UK veteran's mental health charity. Recruitment, consent and data collection is performed automatically through the Drinks:Ration platform. The primary outcome is change in self-reported weekly alcohol consumption between baseline (day 0) and 3-month follow-up (day 84) as measured using the Time-Line Follow back for Alcohol Consumption; secondary outcome measures include 1) change in baseline to 3-month follow-up (day 84) Alcohol Use Disorder Identification Test score, and 2) change in baseline to 3-month follow-up (day 84) World Health Organisation Quality of Life-BREF score to assess Quality of Adjusted Life Years. Process evaluation measures include 1) app usage, and 2) usability ratings as measured by the mHealth App Usability Questionnaire. The primary and secondary outcomes will also be re-assessed at 6-month follow-up (day 168) to assess the longer-term benefits of the intervention and reported as a secondary outcome. The study will begin recruitment in September 2020 and is expected to require 12 months to complete. Study results should be published in 2022.

DETAILED DESCRIPTION:
Alcohol misuse is common in the United Kingdom (UK) Armed Forces (AF), with the prevalence rates higher in the AF than the general population. Research indicates that the trend continues after personnel leave service ('veteran' or 'ex-serving' are used interchangeably in the UK). It has been estimated that more than 50% of those who have left the AF meet the criteria for hazardous alcohol use, a score of eight or above on the Alcohol Use Disorders Identification Test (AUDIT).

The last two decades has seen a proliferation in the use of digital technologies to support brief intervention management and treatment of alcohol misuse in the general public, yet little attention has focused forwards the AF community. In the late 1990's interventions were commonly delivered via a computer using CD-ROM-based programmes, but with the advent of the World Wide Web many new opportunities arose to harness increase reach, provide real-time monitoring, and offer personalised treatment. This includes the use of Short Message Service (SMS) which have been shown to be effective in encouraging people to change their behaviour.

The aim of this Randomised Controlled Trial (RCT) is to assess the efficacy of a 28-day brief alcohol intervention delivered via a smartphone app (Drinks:Ration) in reducing self-reported weekly alcohol consumption between baseline and 3 months (day 84) among veterans who drink at a hazardous or harmful level and are receiving, or have received, support for mental health symptoms in a clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be included if they have downloaded the app onto an iOS or Android device;
* Participants will be included if they are 18 years of age or older;
* Participants will be included if they live in the UK;
* Participants will be included if they consume fourteen units (approximately 140g of alcohol) of alcohol or more per week as measured using Time-Line Follow back for Alcohol Consumption at baseline (day 0);
* Participants will be included if they provide a mobile phone number; and
* Are a veteran of the UK Armed Forces.

Exclusion Criteria:

* Participants will be excluded if they are listed as being 'red' risk by Combat Stress, which is determined by the clinical team following an initial assessment and is based on a traffic light system to assess risk, where red indicates an immediate high risk to the individual and/or others. The application of 'red' risk is applied independently of the research team and is used only where participation in the study could impact clinical treatment. The exclusion will apply only during contact list data extraction.
* Participants will be excluded if they do not have a mobile phone; and
* Participants will be excluded if they have not given Combat Stress consent for contact for research purposes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2022-03-28 (Actual)

PRIMARY OUTCOMES:
Alcohol consumption change | 3 months
  The primary outcome measure is change between self-reported alcohol consumption as measured by the 7-day timeline to Followback over the previous seven days between baseline (day 0) and 3-month follow-up (day 84)

SECONDARY OUTCOMES:
Change in Alcohol Use Disorder Identification Test score | 3 months
  Exploring the change in baseline (day 0) to follow-up (day 84) Alcohol Use Disorder Identification Test score (range between 0-40; 8 or more indicates increased risk)
Change in Quality of Adjusted Life Years | 3 months
  Exploring change in baseline (day 0) to follow-up (day 84) in World Health Organization Quality of Life-BREF questionnaire to assess Quality of Adjusted Life Years (unit measure: life years)

OTHER OUTCOMES:
Repeated measure analysis | 6 months
  The Primary Outcome Measure and Secondary Outcome Measures 2 and Secondary Outcome Measures 3 will be reassessed at month 6. The analysis will explore the difference in alcohol unit consumed (continuous), Alcohol Use Disorder Identification Test score (0-40; a score 8 > indicates increased risk) and the World Health Organization Quality of Life-BREF score (unit measure: life years) between baseline, day 28 (1 month), day 84 (3 months) and 6 months (164 days). The analysis will report change between baseline and each timepoints.
Usage of the Drinks:Ration app | 28-days
  An additional analysis will explore the usage of the app over the first 28 days by participants (in intervention period). This will be reported as the number of app engagements per week (frequency count), the number of pages viewed per week (frequency count) and the number of participants to open the app each week (frequency count - participants).
Evaluating usability of Drinks:Ration | 28-days
  Participants will be asked to complete the mHealth App Usability Questionnaire at day 28, a 16-item, 7-point Likert scale questionnaire focused on assessing the usability of a smartphone app. Each question is focused on a specific domain, the highest the rating (7=excellent) the more positive the outcome. Participants responses will be aggregated per question, and reported as a mean value.

CONTACTS AND LOCATIONS:
Locations (1):
- Combat Stress, Leatherhead, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
To promote open science, consent will be sought from participants to share their data anonymously for research purposes. This data will be released upon completion of the study. Only questionnaire response, remote measurement technology data and alcohol consumption statistics will be shared. All data will be de-identified, and no personal data will be released.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Data is available for access via contact to the lead researcher.
Access Criteria: Researchers will be required to sign a Data Sharing Agreement.
URL: https://drinksration.app/

REFERENCES:
- [Background] Leightley D, Rona RJ, Shearer J, Williamson C, Gunasinghe C, Simms A, Fear NT, Goodwin L, Murphy D. Evaluating the Efficacy of a Mobile App (Drinks:Ration) and Personalized Text and Push Messaging to Reduce Alcohol Consumption in a Veteran Population: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2020 Oct 2;9(10):e19720. doi: 10.2196/19720. PMID 33006569
- [Background] Williamson C, White K, Rona RJ, Simms A, Fear NT, Goodwin L, Murphy D, Leightley D. Smartphone-based alcohol interventions: A systematic review on the role of notifications in changing behaviors toward alcohol. Subst Abus. 2022;43(1):1231-1244. doi: 10.1080/08897077.2022.2074595. PMID 35670777
- [Result] Puddephatt JA, Leightley D, Palmer L, Jones N, Mahmoodi T, Drummond C, Rona RJ, Fear NT, Field M, Goodwin L. A Qualitative Evaluation of the Acceptability of a Tailored Smartphone Alcohol Intervention for a Military Population: Information About Drinking for Ex-Serving Personnel (InDEx) App. JMIR Mhealth Uhealth. 2019 May 24;7(5):e12267. doi: 10.2196/12267. PMID 31127726
- [Result] Leightley D, Puddephatt JA, Jones N, Mahmoodi T, Chui Z, Field M, Drummond C, Rona RJ, Fear NT, Goodwin L. A Smartphone App and Personalized Text Messaging Framework (InDEx) to Monitor and Reduce Alcohol Use in Ex-Serving Personnel: Development and Feasibility Study. JMIR Mhealth Uhealth. 2018 Sep 11;6(9):e10074. doi: 10.2196/10074. PMID 30206054
- [Result] Leightley D, Puddephatt JA, Goodwin L, Rona R, Fear NT. InDEx: Open Source iOS and Android Software for Self-Reporting and Monitoring of Alcohol Consumption. J Open Res Softw. 2018 Mar 23;6:13. doi: 10.5334/jors.207. PMID 29795769
- [Result] Leightley D, Williamson C, Rona RJ, Carr E, Shearer J, Davis JP, Simms A, Fear NT, Goodwin L, Murphy D. Evaluating the Efficacy of the Drinks:Ration Mobile App to Reduce Alcohol Consumption in a Help-Seeking Military Veteran Population: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2022 Jun 20;10(6):e38991. doi: 10.2196/38991. PMID 35724966
- [Derived] Trompeter N, Williamson C, Rona RJ, Carr E, Simms A, Agwuna J, Fear NT, Goodwin L, Murphy D, Shearer J, Leightley D. Shorter communications: Exploring the impact of a brief smartphone-based alcohol intervention app (DrinksRation) on the quality of life of UK military veterans. Behav Res Ther. 2024 Jun;177:104540. doi: 10.1016/j.brat.2024.104540. Epub 2024 Apr 6. PMID 38598898
- See also: Drinks:Ration website — https://drinksration.app/